CLINICAL TRIAL: NCT04215185
Title: Prospective Open Study for the Development of CS6BP Continuous, Absolute, Non-Inflating Measurement of Blood Pressure
Brief Title: Data Collection of BP Values by CS6BP
Acronym: BPI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CardiacSense Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 004_BPI_DC_OS
Record Dates: First submitted 2019-12-23; First posted 2020-01-02 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Blood Pressure
MeSH Terms: interventions — Vascular Access Devices

STUDY DESIGN:
Intervention Model Description: Non-anaesthetized subjects in the ICU (Intensive Care Unit) or in the CICU (Cardiac Intensive Care Unit) with arterial line placement in the radial artery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Blood pressure monitor (Experimental): The CS6BP device will be placed on non-anesthetized subjects in the ICU (Intensive Care Unit) with arterial line placement in the radial artery. The first measurement will be for up to 24h; subsequent measures will be up to 5h.
  Interventions: Device: Arterial LIne

INTERVENTIONS:
Device: Arterial LIne — Continuous non-invasive recording of CS6BP will be taken parallel to the recording of an invasive arterial line. ECG data recorded in the ICU will also be collected.
  Other Names: A-Line

SUMMARY:
The primary objective of this research is to collect data to develop an algorithm for continuous, non-inflating measurement of absolute, long-term Blood Pressure using the CS6BP device and to evaluate the safety of the CS6BP.

DETAILED DESCRIPTION:
The study will take place in the ICU (Intensive Care Unit) on non-anesthetized subjects with an arterial line inserted into the radial artery. The CS6BP non-invasive continuous recording will be collected parallel to an invasive arterial line recording. ECG data that was recorded in the ICU will be collected as well.

The study will include up to 80 subjects.

The subject may be measured by the CS6BP device more than once to check reproducibility. The first measurement may take up to 24h; Subsequent measurements may take up to 5h. All the data analysis will be done offline.

ELIGIBILITY:
Inclusion Criteria:

* Age of eighteen (18) year and above
* Ability and willingness to sign an informed consent form
* Monitored by radial arterial line

Exclusion Criteria:

* Subjects with hemodynamic support
* Subjects receiving more than 2-3 l of fluid per 24h
* Subjects with septic shock
* Subjects with distal edema
* Subjects with arms trauma, where the watch is not wearable
* Subjects where the radial artery could not be palpate
* Subjects with life expectancy of less than 24h.
* Subjects who are currently enrolled in another clinical investigation in which the intervention might compromise the safety of the subject's participation in this study
* Any concomitant condition which, in the opinion of the investigator, would not allow safe participation in the study (e.g. drug addiction, alcohol abuse, emotional/psychological diagnosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-07-03 (Actual); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
Safety of CardiacSense 1BP: Incidence and severity of device related Adverse Events | measurement time (up to 24 hours)
  Incidence and severity of device related Adverse Events
Collection of data from CardicacSense1BP measurements for algorithm development | measurement time (up to 24 hours)
  CardicacSense1BP data will be collected in parallel with blood pressure data from ICU a- line .

CONTACTS AND LOCATIONS:
Overall Officials: Adi Nimrod, MD, Principal Investigator — Director Intensive Care Unit, Tel-Aviv Sourasky Medical Center
Locations (1):
- Sourasky Medical Center, Tel Aviv, Israel